CLINICAL TRIAL: NCT04155554
Title: The Effects of Switching From Dolutegravir/Lamivudine/Abacavir (d/l/a) to Bictegravir/Emtricitabine/Tenofovir Alafenamide (b/f/Taf) in Patients With Suppressed Viral Load on Neuropsychiatric Side Effects and Neurocognitive Function
Brief Title: Neurological Monitoring in Patients Switching From Dolutegravir Based Regimen to Bictegravir Based Regimen
Acronym: DOBINeuro
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Senese (Other)
Collaborators: Catholic University of the Sacred Heart (Other); Ospedale Policlinico San Martino (Other); Azienda Ospedaliera San Paolo (Other); Ospedale Amedeo di Savoia (Other)
Responsible Party: Principal Investigator, Barbara Rossetti, Principal Investigator, Azienda Ospedaliera Universitaria Senese
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-004885-32
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: HIV-1-infection
Keywords: HIV; Neurocognitive functions; Neuropsychiatric side effects; Bictegravir; INSTI
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination; abacavir, dolutegravir, and lamivudine drug combination

STUDY DESIGN:
Intervention Model Description: Prospective, randomized study (1: 1), open-label, controlled, phase 3, multicenter, non-profit
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bictegravir/emtricitabine/tenofovir alafenamide (Experimental): Patients with suppressed viral load switching from dolutegravur/lamivudina/abacavir (50/300/600 mg) 1 tablet OD to bictegravir/emtricitabine/tenofovir alafenamide (50/200/25 mg) 1 tablet OD
  Interventions: Drug: Bictegravir/emtricitabine/tenofovir alafenamide
- Dolutegravir/lamivudine/abacavir (Active Comparator): Patients with suppressed viral load continuing dolutegravir/lamivudine/abacavir (50/300/600 mg) 1 tablet OD
  Interventions: Drug: Dolutegravir/lamivudine/abacavir

INTERVENTIONS:
Drug: Bictegravir/emtricitabine/tenofovir alafenamide — Switch patients from dolutegravir/lamivudine/abacavir to bictegravir/emtricitabine/tenefovir alafenamide to study neuropsychiatric side effects and neurocognitive function
  Other Names: Biktarvy
  Arms: Bictegravir/emtricitabine/tenofovir alafenamide
Drug: Dolutegravir/lamivudine/abacavir — Continuing dolutegravir/lamivudine/abacavir to study neuropsychiatric side effects and neurocognitive function
  Other Names: Triumeq
  Arms: Dolutegravir/lamivudine/abacavir

SUMMARY:
Prospective, randomized study (1: 1), open-label, controlled, phase 3, multicenter, non-profit. The hypothesis of the present study is that bictegravir is associated with a lower incidence and severity of neuropsychiatric symptoms than dolutegravir.

DETAILED DESCRIPTION:
Prospective, randomized study (1: 1), open-label, controlled, phase 3, multicenter, non-profit. The hypothesis of the present study is that bictegravir is associated with a lower incidence and severity of neuropsychiatric symptoms than dolutegravir. The main outcome measure will be a global severity index (GSI) of neuropsychiatric symptoms arising from 10 symptom domains, including somatization, obsessive-compulsiveness, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism. The secondary outcomes are to compare, between arms and during follow up, neuropsychiatric symptoms severity, neurocognitive performance, changes in self-reported symptoms, adherence and HR-QoL, correlation between symptoms (neuropsychiatric and other), drug exposure and HR-QoL, proportion of adverse events, proportion of virological failures and antiretrovirals resistance at virological failure.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* HIV-1 infection
* HIV RNA <50 copies/mL >12 months (including patients with 1 blip 50-200 cp/mL before screening, not confirmed)
* On treatment with dolutegravir/abacavir/lamivudine >6 months

Exclusion Criteria:

* Previous AIDS events
* Pregnancy or pregnancy plan
* Decompensated cirrhosis (B or C CPT status)
* Intake of alcohol, substances, other drugs that may affect neurocognitive performances
* Necessity to receive drugs that may require dosing adjustment of dolutegravir or bictegravir
* Certified diagnosis of major depression, psychosis, history of suicidal attempts
* Treatment with antidepressants or antipsychotic drugs
* History of virological failure with INSTIs
* Lack of knowledge of italian language
* Impossibility to obtain informed written consent
* HBsAg positivity
* Estimated glomerular filtration rate by CK-EPI <50 mL/min per 1.73 m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
neuropsychiatric symptoms severity in 3 months | 3 months
  change in neuropsychiatric symptoms severity, using the Symptom Checklist-90-R, 3 months after switching to bictegravir or continuing dolutegravir (on treatment analysis).

SECONDARY OUTCOMES:
neuropsychiatric symptoms severity in 3 and 12 months | 12 months
  change in neuropsychiatric symptoms severity, each of the 10 symptoms analyzed separately using the Symptom Checklist-90-R, 3 and 12 months after switching to bictegravir or dolutegravir (on treatment analysis)
Mini International Neuropsychiatric Interview Plus subscale for suicide risk | 12 months
  change in neuropsychiatric symptoms severity, using the Mini International Neuropsychiatric Interview Plus subscale for suicide risk, 3 and 12 months after switching to bictegravir or dolutegravir (on treatment analysis). Suicide risk (five questions, score range 0-33 points) in the last 30 days was classified as low (1-5), moderate (6-9), or high (10).
neurocognitive performance | 12 months
  change in neurocognitive performance, using a comprehensive and validated neuropsychological battery, 12 months after switching to bictegravir or dolutegravir (on treatment analysis).
  The neurocognitive performance is calculated by averaging the individual deficit scores from each neurocognitive test. Deficit scores for each test were calculated from age-, education-, -adjusted raw scores.
neurocognitive impairment and neuropsychiatric symptoms | 12 months
  comparison of the inter-arm and intra-arm incidence of neurocognitive impairment (on the basis of Frascati criteria) at 12 months and neuropsychiatric symptoms (using the Symptom Checklist-90-R) at 3 (on treatment analysis) and 12 months (ITT-exposed, using LOCF)
self-reported symptoms (21 items, 0-5 points for each), adherence (0-100%) and HR-QoL (9 items, 0-5 points for each) | 12 months
  changes in self-reported symptoms, adherence and HR-QoL (using validated questionnaires) during the first year of follow up (ITT-exposed, using LOCF).
drug exposure | 12 months
  correlation between symptoms (neuropsychiatric and other), drug exposure and HR-QoL during the first year of follow up (ITT-exposed, using LOCF).
adverse events | 12 months
  proportion of adverse events and serious adverse events and of patients discontinuing due to side effects in both arms
virological failures | 12 months
  proportion of virological failures and antiretrovirals resistance at virological failure
Treatment Satisfaction | 12 months
  change in Treatment Satisfaction between arms as per specific questionnaire (TSQM Version 1.4, 15 questions, from 0 to 79 points as maximum)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Rossetti, PhD, Principal Investigator — Azienda Ospedaliera Universitaria Senese
Locations (1):
- Barbara Rossetti, Siena, Italy

IPD SHARING:
Plan to Share IPD: No